CLINICAL TRIAL: NCT00581984
Title: McGhan Medical Silicone-Filled Breast Implant Adjunct Study
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 98-089
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Breast Reconstruction With Silicone Implants
Keywords: breast cancer; breast reconstruction; silicone implants
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
This study will collect 5 year data about any possible health problems associated with breast implants. This data will be used to help see if the implants are both safe and effective. If they are proven safe and effective, they will continue to be available. If they are not proven safe and effective to the satisfaction of the FDA, they may not be available in the future.

DETAILED DESCRIPTION:
This prospective clinical study is being undertaken to document the safety of McGhan Medical Silicone-Filled Breast Implants. Patients will be evaluated pre-operatively, intraoperatively, and at one, three and five years following implant surgery. Safety of McGhan Medical Silicone-Filled Breast Implants will be assessed based on the incidence of medical complications, implant failure and serious adverse effects.

This prospective clinical study of McGhan Medical Silicone-Filled Breast Implants is part of an ongoing research effort to document the safety and effectiveness of silicone-filled breast implants.

ELIGIBILITY:
Inclusion Criteria:

* Females of any age for which breast reconstruction is considered appropriate. (Patients under 18 years old require parental/legal guardian consent to participate).
* Have any of the following conditions or situations present:

  * Post mastectomy surgical removal of the breast for cancer or other diseases;
  * Post trauma or post surgery where there was total or partial removal of the breast resulting in significant deformity.(for any reason);
  * Severe ptosis requiring reconstruction (i.e. mastopexy);.
  * Any congenital or acquired discrepancy in breast size such as to represent a significant physical deformity. This does not include normal variants of asymmetry. Examples include, but are not limited to:Pectus excavatum, Pectus carinatum; Thoracic hypoplasia (Poland's syndrome, Scoliosis; Isolated rib deformities; Tuberous breasts; Congenital absence
  * Revision of implant procedure due to any of the following circumstances;
* Previous augmentation or reconstruction with silicone- or saline-filled implants where problems exist, such as implant. rapture or significant capsular contracture (Baker Grade III or IV) requiring revision;

  * Contralateral mammaplasty in unaffected breast as a result of the affected breast requiring surgery (for one of the aforementioned circumstances), when medically indicated to provide symmetry.
* Adequate tissue available to cover implants.
* Saline-filled implants are not an appropriate choice.
* Willingness to follow all study requirements, such as agreeing to all required follow-up visits, and acceptance of the risks involved as indicated by signing of the Patient Informed Consent document.

Exclusion Criteria:

* Advanced fibrocystic disease considered to be premalignant-without accompanying subcutaneous mastectomy.
* Existing carcinoma of the breast, without mastectomy.
* Abscess or infection in the body at the time of enrollment.
* Pregnant or nursing.
* Have any disease, including uncontrolled diabetes; which is clinically known to impact wound healing ability.
* Show tissue characteristics which are clinically incompatible with mammaplasty, such as tissue damage resulting from radiation, inadequate tissue, compromised vascularity or ulceration.
* Have, or under treatment for, any condition which, in the opinion of the surgeon, may constitute an unwarranted surgical risk.
* Show psychological characteristics which, in the opinion of the surgeon, may be incompatible with the surgical procedure and the prosthesis, such as inappropriate attitude or motivation.
* Wish to have augmentation mammaplasty, but do not have at least one of the diagnoses identified in Patient Inclusion Criteria item G #2, pages 7 & 8.
* Are not willing to undergo further surgery for revision, if medically required.
* Diagnosis of lupus or scleroderma.
* Replacement of saline-filled implants solely for a less than desirable cosmetic outcome, such as wrinkling.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Females who are candidates for breast reconstructio
Sampling Method: Non-Probability Sample
Enrollment: 1016 (Actual)
Dates: Start 1998-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Evidence of breast implant complications | 10 years 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Cordeiro, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org